CLINICAL TRIAL: NCT06423287
Title: Effects of Time-Restricted Eating With Lactobacillus Plantarum LP-KFY04 Supplementation on Overweight / Obese Individuals : A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effects of TRE With Lactobacillus Plantarum LP-KFY04 Supplementation on Overweight / Obese Individuals
Acronym: TRELO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024LX0016_GY
Record Dates: First submitted 2024-04-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Obesity; Time-restricted Diet; Probiotic Compound LP-KFY04; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum LP-KFY04 (Experimental): Patients in the treatment group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of Lactobacillus plantarum LP-KFY04 over 12 weeks' trial.
  Interventions: Dietary Supplement: Lactobacillus plantarum LP-KFY04
- placebo (Placebo Comparator): Patients in the control group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of placebo over 12 weeks' trial.
  Interventions: Other: Take placebo in addition to the limited diet.

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum LP-KFY04 — Patients in the treatment group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of Lactobacillus plantarum LP-KFY04 over 12 weeks' trial.
  Arms: Lactobacillus plantarum LP-KFY04
Other: Take placebo in addition to the limited diet. — Patients in the control group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of placebo over 12 weeks'trial.
  Arms: placebo

SUMMARY:
With the improvement of the quality of life, multi-nutritional dietary intake today has provided people with a solid foundation for their health profiles. Time-restricted eating is found to be an effective method to prevent and control obesity, helping obese patients to lose weight in a way of reshaping the gut microbiota. Regulation of gut microbiota, as a valid weight-loss strategy, can be achieved by oral supplementation of probiotics. This study aims to evaluate the effectiveness of time-restricted eating combined with Lactobacillus Plantarum LP-KFY04 on overweight/obese population through a multi-center, randomized and double-blind clinical trial.

DETAILED DESCRIPTION:
With the improvement of the quality of life, multi-nutritional dietary intake today has provided people with a solid foundation for their health profiles. Time-restricted eating is found to be an effective method to prevent and control obesity, helping obese patients to lose weight in a way of reshaping the gut microbiota. Regulation of gut microbiota, as a valid weight-loss strategy, can be achieved by oral supplementation of probiotics. This study aims to evaluate the effectiveness of time-restricted eating combined with Lactobacillus Plantarum LP-KFY04 on overweight/obese population through a multi-center, randomized and double-blind clinical trial.Patients in the treatment group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of Lactobacillus plantarum LP-KFY04 over 12 weeks'trial.Patients in the control group will be instructed to eat in an 8-hour time window (a set period of time decided by the patients) with supplementation of placebo over 12 weeks' trial.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 65 years old
2. BMI 24.0 to 40kg/m2
3. Patients who are aware of the purpose of the trail, willing to participate in the trial and sign informed consent forms, and comply with all requirements (including those during follow-up and evaluation investigations)

Exclusion Criteria:

1. History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis;
2. Diagnosis of type 1 or type 2 diabetes and prescribing hypoglycemic therapy
3. History of malignant tumors
4. Serious liver dysfunction or chronic kidney disease (aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2)
5. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction, or stroke) within the past 6 months
6. History of serious gastrointestinal disease or gastrointestinal surgery within the past 12 months
7. History of Cushing's syndrome, hypothyroidism, acromegaly, and hypothalamic obesity
8. Smoking or have smoked within the past 3 months of the screening period
9. Drinking alcohol or drinking more than 15 grams of alcohol per day within the past 3 months of the screening period
10. Taking any medicine that may affect weight or metabolism within the past 6 months, including weight loss medications, antipsychotics, or other medications identified by the researchers
11. Currently involving in a weight loss program or having significant weight change within the past 3 months (> 5% of current weight)
12. Women who are pregnant or planning for pregnant
13. Patients who are unable to complete 12-week follow-up (due to health conditions or immigration reasons)
14. Patients who are unwilling or unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of body weight from baseline to 12 weeks after intervention | 12 weeks

SECONDARY OUTCOMES:
Changes of BMI compared with baseline in subjects | 12 weeks
Changes of waist circumference compared with baseline in subjects | 12 weeks
Changes of body fat percentage (BF%) compared with baseline assessed by dual-energy X-ray absorptiometry (DEXA) | 12 weeks
Change of subjects' HOMA-IR compared with baseline | 12 weeks
Changes of blood pressure in subjects compared with baseline | 12 weeks
Changes of blood glucose in subjects compared with baseline | 12 weeks
Changes of blood lipids in subjects compared with baseline | 12 weeks
  Blood lipids includes total cholesterol、triglyceride、LDL-c、HDL-c.
Changes of intestinal microbial composition compared with baseline in subjects | 12 weeks
  Species of intestinal microbial includes Firmicutes、Bacteroidetes、Proteobacteria、Actinobacteriota、Verrucomicrobia、Fusobacteria.
Changes of intestinal microbial abundance compared with baseline in subjects | 12 weeks
  Proportion of intestinal microbial such as Firmicutes、Bacteroidetes、Proteobacteria、Actinobacteriota、Verrucomicrobia、Fusobacteria
Changes of plasma metabolite compared with baseline in subjects | 12 weeks
  Plasma metabolite includes arachidonic acid 、betaine、glutathione and so on.
The incidence of adverse events in two groups of subjects | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chen, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China